CLINICAL TRIAL: NCT02045719
Title: Phase II Clinical Trial of Uncaria Tomentosa (Cat´s Claw) in Patients With Advanced Solid Tumors
Acronym: cat´sclaw
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Faculdade de Medicina do ABC (Other)
Responsible Party: Principal Investigator, Felipe Melo Cruz, MsC, Faculdade de Medicina do ABC
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ABC2013
Record Dates: First submitted 2014-01-23; First posted 2014-01-27 (Estimated); Last update posted 2014-01-27 (Estimated); Status verified 2014-01

CONDITIONS: Solid Tumors
Keywords: cat´s claw; uncaria tomentosa; quality of life; no further therapeutic options
MeSH Terms: interventions — cat's claw extract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- cat's claw (Experimental): 100 mg dose of a dry extract of U. tomentosa three times per day
  Interventions: Drug: uncaria tomentosa (cat´s claw)

INTERVENTIONS:
Drug: uncaria tomentosa (cat´s claw)
  Other Names: 100 mg dose of a dry extract of U. tomentosa three times per day

SUMMARY:
Cat's claw (Uncaria tomentosa) is a native amazonic plant that exhibits anti-inflammatory and antitumor properties. Patients and methods: This prospective phase II study will assess the effects of a 100-mg dose of a dry extract of U. tomentosa three times per day on individuals with advanced solid tumors, with no further therapeutic options and with at least 2 months life expectancy. In addition, several biochemical and inflammatory parameters will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* individuals with advanced solid tumors, with no further therapeutic options and with at least 2 moths life expectancy
* individuals 18 years of age and older
* creatinine levels up to twice the upper limit of normal (ULN)
* alanine (ALT) and aspartate (ASP) transaminase levels up to twice the ULN and direct bilirubin (DB) levels up to 1.5 times the ULN
* in cases with pre-existing liver disease, the ALT, ASP and DB levels could be up to 2.5 times the ULN

Exclusion Criteria:

* pregnant and breastfeeding women
* individuals using chemotherapy or other tumor-targeting antineoplastic treatments, except for antalgic radiotherapy
* severe kidney or liver failure
* known hypersensitiveness to the components of the medication used
* past history of emotional disorders that could interfere with the data collection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2013-12; Primary Completion 2014-07 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
assessment of benefits on quality of life after treatment during two months | two months
  Assess the efficacy and safety of a dry extract of U. tomentosa on individuals who had solid tumors with no further therapeutic options

CONTACTS AND LOCATIONS:
Locations (1):
- Centro de Estudos e Pesquisa em Hematologia e Oncologia, Santo André, São Paulo, Brazil